CLINICAL TRIAL: NCT05862649
Title: A Multicenter Longitudinal Study to Evaluate the Correlation Between Oculometric Measures and Clinical Assessment in Patients With Idiopathic Parkinson's Disease (PALOMA Trial)
Brief Title: Evaluation of Correlation Between Oculometric Measures and Clinical Assessment in Parkinson's Disease
Acronym: PALOMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NeuraLight (Industry)
Collaborators: European Clinical Research Infrastructure Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL/PD/2023-1
Record Dates: First submitted 2023-05-08; First posted 2023-05-17 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD patients (Experimental): Men and women with idiopathic PD (Hoehn & Yahr scale 1-2) aged 40-85 years
  Interventions: Other: NeuraLight

INTERVENTIONS:
Other: NeuraLight — NeuraLight software-based platform

SUMMARY:
This is a multicenter longitudinal study in about 300 patients with Idiopathic Parkinson's disease, who will be evaluated in several clinical centers with a clinical assessment and an oculometric examination during a time period with specific intervals. This study aims to evaluate the correlation between oculometric measures and clinical assessment over time, as well as the potential to detect early change in clinical status using an oculometric assessment.

DETAILED DESCRIPTION:
This is an multicenter longitudinal study, in about 300 patients with idiopathic PD in several centers. The aim of this study is to evaluate the correlations between oculometric measures and clinical assessment, e.g. the Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) and the MoCA score over time ,in subjects who meet the inclusion and exclusion criteria, and who provide a signed Informed Consent. In addition, the investigators aim to demonstrate that oculometric measures are able to detect patient deterioration faster than can be detected using the currently available clinical assessment tools. All patients will be assessed over a period of 12 months (5 assessments, at 0, 3, 6, 9, 12 months). During this time period, every subject who consents will undergo a NeuraLight session including oculometric measurements and eye-tracking recordings using a novel software-based platform and an eye- tracking system (Tobii, CE-marked class B approved device) (approx. 30 minutes). The oculometric evaluation will occur for every patient every 3 months. All assessments will be performed during a clinic visit unless authorized to be conducted remotely. During the study, the sponsor will be blinded to the private details of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with idiopathic PD (Hoehn & Yahr scale 1-2)
* Age between 40 and 85 years old
* 0 to 5 years' time since diagnosis
* Normal or corrected vision
* Ability to follow instructions
* Willing and able to sign an informed consent form
* No anticipated changes in PD medications from baseline throughout the study duration based on clinical status during screening
* If treated, stable on treatment for at least 3 months

Exclusion Criteria:

* Inability to sit for 40 minutes on a chair in a calm manner
* Personal or 1st degree relative history of epilepsy
* Additional neurological diseases
* Drug or alcohol abuse (except for using medical cannabis during 24 hours prior NL examination date)
* Pregnancy or a potential pregnancy (self-declaration)

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Change of saccadic latency over time as evaluated during visits | 12 months
  Difference between saccadic latency (ms) as quantified during each visit by the NeuraLight test measured using a statistical comparison of values (e.g. t-test, ANOVA), p>0.05) over time during study period
Change of anti-saccadic error rates over time as evaluated during visits | 12 months
  Difference between anti-saccadic error rates (%) as quantified during each visit by the NeuraLight test measured using a statistical comparison of values (e.g. t-test, ANOVA), p>0.05) over time during study period
Change of smooth pursuit speed over time as evaluated during visits | 12 months
  Difference between smooth pursuit speed (ms)as quantified during each visit by the NeuraLight test measured using a statistical comparison of values (e.g. t-test, ANOVA), p>0.05) over time during study period
Correlation between MDS-UPDRS score and its parts with saccadic latency | 12 months
  The correlation between the Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS, scored 0-to a maximum total of 199, indicating the worst possible disability from PD) and its parts with saccadic latency (ms) measured using R-Square (high correlation>0.5, moderate correlation 0.2-0.5, low correlation<0.2), p<0.05) according to MDS-UPDRS scores at visits
Correlation between MDS-UPDRS score and its parts with anti-saccadic error rates | 12 months
  The correlation between Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS, scored 0-to a maximum total of 199, indicating the worst possible disability from PD) and its parts with anti-saccadic error rates (%), measured using R-Square (high correlation>0.5, moderate correlation 0.2-0.5, low correlation<0.2), p<0.05) according to the MDS-UPDRS scores at visits
Correlation between MDS-UPDRS score and its parts with smooth pursuit | 12 months
  The correlation between Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS, scored 0-to a maximum total of 199, indicating the worst possible disability from PD) and its parts with smooth pursuit speed (ms) measured using R-Square (high correlation>0.5, moderate correlation 0.2-0.5, low correlation<0.2), p<0.05) according to the Movement Disorder Society-Sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) at visits

SECONDARY OUTCOMES:
Correlation between MoCA score and its parts with saccadic latency | 12 months
  The correlation between MoCA score and its parts with saccadic latency (ms) measured using R-Square (high correlation>0.5, moderate correlation
Correlation between MoCA score and its parts with anti-saccadic error rates | 12 months
  The correlation between the Montreal Cognitive Assessment (MoCA, scored 0- to a total possible score is 30 points, where a score of 26 or above is considered normal) with anti-saccadic error rates (%), measured using R-Square (high correlation>0.5, moderate correlation 0.2-0.5, low correlation<0.2), p<0.05) according to the Montreal Cognitive Assessment (MoCA) at visits
Correlation between MoCA score and its parts with smooth pursuit | 12 months
  The correlation between Montreal Cognitive Assessment (MoCA, scored 0- to a total possible score is 30 points, where a score of 26 or above is considered normal) with smooth pursuit speed (ms) measured using R-Square (high correlation>0.5, moderate correlation 0.2-0.5, low correlation<0.2), p<0.05) according to the Montreal Cognitive Assessment (MoCA) at visits
Using the retrieved data of collected NeuraLight oculometric measures for calibration of prediction models of MDS-UPDRS clinical endpoint | 12 months
  Optimization of a feature selection model (Fisher's Linear Discriminant Analysis (LDA)) on NeuraLight oculometric measures used for a logistic regression model of Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating ScaleMDS-UPDRS, scored 0-to a maximum total of 199, indicating the worst possible disability from PD) and its parts with a relative root mean square error (RMSE) of <0.1
Using the retrieved data of collected NeuraLight oculometric measures for calibration of prediction models of MoCA clinical endpoint | 12 months
  Optimization of a feature selection model (Fisher's Linear Discriminant Analysis (LDA)) on NeuraLight oculometric measures used for a logistic regression model of Montreal Cognitive Assessment (MoCA, scored 0- to a total possible score is 30 points, where a score of 26 or above is considered normal) with a relative root mean square error (RMSE) of <0.1

CONTACTS AND LOCATIONS:
Overall Officials: Christina Januário, MD, Principal Investigator — University of Coimbra; Richard Armstrong, MD, Principal Investigator — The VCTC; Pablo Mir, MD, Principal Investigator — Instituto de Biomedicina de Sevilla (IBiS; Michelle Tosin, PhD, Principal Investigator — Rush Medical University Center; Bettina Balint, MD, Principal Investigator — University Hospital, Zürich
Locations (5):
- Rush University, Chicago, Illinois, United States
- AIBILI research center, Coimbra, Portugal
- Instituto de Biomedicina de Sevilla (IBiS), Seville, Spain
- University Hospital Zürich, Zurich, Switzerland
- The VCTC, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No